CLINICAL TRIAL: NCT02009748
Title: Vitamin D Supplementation in Cirrhotic Patients: A Randomized, Multi-center, Double-blind, Placebo Controlled Trial to Evaluate Vitamin D Supplementation on Serum 25-hydroxyvitamin D Levels in Cirrhotic Patients
Brief Title: Vitamin D Supplementation in Cirrhotic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Rudolf Stauber, MD, Univ. Prof. Dr. med., Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VITDZIRR
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Cirrhosis; Vitamin D Deficiency
MeSH Terms: conditions — Fibrosis; Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D supplementation (Active Comparator): Colecalciferol 2.800 IU/day
  Interventions: Dietary Supplement: Vitamin D supplementation
- Placebo (Placebo Comparator): Vehicle (coconut oil)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D supplementation — oral administration of colecalciferol 2.800 IU once daily
  Arms: Vitamin D supplementation
Dietary Supplement: Placebo — oral administration of placebo (vehicle) once daily
  Arms: Placebo

SUMMARY:
Previous studies suggested that vitamin D deficiency is highly prevalent in cirrhotic patients and is related to the degree of liver dysfunction as well as mortality. In gastrointestinal disorders, vitamin D absorption can be highly reduced.

We herein aim to investigate the efficacy of oral vitamin D supplementation in cirrhotic patients with vitamin D insufficiency.

DETAILED DESCRIPTION:
Cirrhosis of the liver is a slowly progressive disease with a high number of complications like hepatic encephalopathy, gastrointestinal bleeding, ascites, renal failure and hepatocellular cancer leading to death. Cirrhosis as a cause of death has increased progressively in the mortality data for the general population.

This terminal liver disease as a complication of chronic viral hepatitis, alcoholism and metabolic disorders, with genetic and non-genetic predisposition, may be linked to nutritional aberration as a precursor to or an effect of the illness. Previous studies suggested that chronic liver diseases may be related to high prevalence of vitamin D deficiency and in gastrointestinal disorders the vitamin D absorption can be highly reduced.

Patients with cirrhosis are often presented with malnutrition and one of the limiting factors of the intestinal malabsorption is the portal hypertension due to the liver disease. Beside nutrition the main source of vitamin D is sunlight and ultraviolet-B inducing the conversion of 7-dehydrocholesterol to vitamin D in the skin; therefore limited sunlight exposure of the skin may lead to an inadequate vitamin D status.

Vitamin D itself is biologically inactive and has to be hydroxylated in the liver to 25-hydroxyvitamin D (25(OH)D) as the main circulating metabolite used for classification of the vitamin D status. 1,25 hydroxyvitamin D (1,25(OH)D) is produced through conversion by the enzyme 1-alpha-hydroxylase in the kidney. This vitamin D metabolite shows a higher affinity for the vitamin D receptor (VDR) compared to 25(OH)D. After binding and activation of the VDR three percent of the human genome will be regulated. Among the main role of vitamin D metabolites to regulate calcium and bone homeostasis, they also show non-skeletal effects with relevance in the development of several chronic diseases. In this context, vitamin D deficiency has been associated with an increased risk of cancer , cardiovascular, autoimmune, and infectious diseases, Based on these findings, a significantly reduced risk of mortality was shown in patients with oral vitamin D supplementation in randomized controlled studies.

Our previously published study presented a prospective association of vitamin D levels with occurrence of hepatic decompensation. Furthermore vitamin D deficiency was associated with high mortality in cirrhotic patients dependent on liver dysfunction. Concerning this aspect the main point is to investigate in this study whether low vitamin D status is the consequence of increasing deterioration of the liver synthesis or may even contribute to liver dysfunction. Low synthesis of vitamin D in the skin can be the result of reduced sunlight exposure and malnutrition and/or malabsorption in cirrhotic patients. On the other hand, organ dysfunction may impair the activity of 25-hydroxylase in the liver. Despite the above mentioned correlation between vitamin D deficiency and liver dysfunction there is still insufficient evidence to recommend oral vitamin D supplementation as a concomitant therapy in clinical practice because there exists no adequately designed randomized controlled trial that evaluates the necessary daily oral dose on vitamin D.

We aim to address this issue in the present study so that the findings of our study will lead to implementation of treatment strategies for maintaining a sufficient vitamin D status in cirrhotic patients.

ELIGIBILITY:
Inclusion Criteria:

* 25(OH)D levels below 30 ng/ml (measured at the baseline visit)
* Compensated and decompensated cirrhosis diagnosed by the hepatologist for at last three months prior to study start
* Age between 18 and 75 years
* Written informed consent
* Negative pregnancy test in women of childbearing potential

Exclusion Criteria:

* Hypercalcemia defined as total serum calcium >2.65 mmol/L
* Pregnancy or lactating women
* Drug intake as part of another clinical study
* Glomerular filtration rate (GFR) < 15 ml/min/1.73m²
* Any disease with an estimated life expectancy below 1 year
* Any clinically significant acute disease requiring drug treatment
* Anticipated chemotherapy or radiation therapy during the study
* Regular intake of more than 800 International Units (IU) of vitamin D during the last 4 weeks before study entry

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-12; Primary Completion 2014-08 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
serum 25(OH)D | 8 weeks after study start

SECONDARY OUTCOMES:
Liver function tests | 8 weeks after study start
  Albumin, prothrombin time, bilirubin
Hyaluronic acid | 8 weeks after study start

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf E Stauber, MD, Principal Investigator — Dept of Internal Medicine, Medical University of Graz
Locations (2):
- Austria (2):
  - Department of Internal Medicine, LKH Hoergas, Gratwein, Styria
  - Department of Internal Medicine, Medical University of Graz, Graz, Styria